CLINICAL TRIAL: NCT00995891
Title: Collection of Blood, Bone Marrow, Skin Biopsies and Buccal Mucosa Samples From Healthy Volunteers for Center for Human Immunology, Autoimmunity, and Inflammatory Diseases (CHI) Protocols Laboratory Research Studies
Brief Title: Collection of Blood, Bone Marrow, and Buccal Mucosa Samples From Healthy Volunteers for Center for Human Immunology, Autoimmunity, and Inflammatory Diseases (CHI) Laboratory Research Studies
Status: Completed | Type: Observational
Sponsor: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Responsible Party: Sponsor
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Other Study IDs: 090229; 09-H-0229
Record Dates: First submitted 2009-10-14; First posted 2009-10-15 (Estimated); Last update posted 2019-12-05 (Actual); Status verified 2018-09-05

CONDITIONS: Healthy Volunteers
Keywords: Laboratory Research Specimens; Biologic Samples; Sample Collection; Tissue Procurement; HV; Healthy Volunteer

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective

SUMMARY:
Background:

- Laboratory research studies require control samples from healthy volunteers to compare with samples from patients. These studies will help researchers better understand and refine treatments for immune system and inflammatory diseases.

Objective:

- To obtain blood, urine, buccal (mouth) mucosa, normal tissue and bone marrow samples and/or leukopheresis cells from healthy volunteers.

Eligibility:

- Healthy individuals at least 8 years of age.

Design:

* Volunteers will be recruited through the Program for Healthy Volunteers, Patient Recruitment and Public Liaison Office, or self-referral through the clinicaltrials.gov Web site.
* Health will be confirmed by a brief history and physical examination and blood work.
* Volunteers 8 years of age and older will provide blood and urine samples using standard procedures. Buccal mucosa samples will be obtained by scraping the insides of both cheeks with a sterile nylon brush.
* Bone marrow samples will be obtained from volunteers 18 years of age and older by taking two aspirates from the posterior iliac crest (an area near the hip).
* Normal tissue samples will be obtained from volunteers 18 years of age and older by taking superficial skin samples (punch biopsies)
* Leukopheresis or lymphapheresis will be performed on volunteers 18 years of age and older to obtain white blood cells for research
* Samples will be assigned a unique code and will be stored until they are no longer of scientific value or the volunteer withdraws consent for their use.

DETAILED DESCRIPTION:
The purpose of this protocol is to collect blood (ages 8 and older), urine (ages 8 and older), buccal mucosa samples (ages 8 and older), normal tissue (ages18 and older) bone marrow (ages 18 and older) and/or leukapheresis cells (ages 18 and older) from healthy volunteers, including pregnant women (ages 18 and older, blood and/or buccal mucosa only). To be enrolled on this study, pregnant women must not carry the diagnosis of an immune-mediated or inflammatory disease, or have signs or symptoms of an immune or inflammatory disease; otherwise they may be eligible for participation on CHI protocol 10-H-0162 in the affected adult cohort. Samples will be used as controls for clinical and translational research in the Center for Human Immunology, Autoimmunity, and Inflammatory Diseases (CHI). These control samples are indispensable for many of our laboratory research projects, including understanding the pathophysiology of a wide variety of immune-mediated and inflammatory diseases.

The primary objective is to provide a mechanism for collection, tracking, storing, dispensing, analyzing and disposing of these laboratory research samples from healthy volunteers.

There is no primary endpoint.

ELIGIBILITY:
* INCLUSION CRITERIA:
* Healthy volunteer (health status confirmed by brief History and Physical Exam and blood work)
* Age 8 years and older (no upper limit) for blood, urine, and buccal mucosa sampling

Or

Ages 18 years or older (no upper limit) for bone marrow or normal tissue sampling and/or leukapheresis cells

Or

Pregnant women (health status confirmed by brief History and Physical Exam and blood work) must be 18 years or older (no upper limit) for blood and/or buccal mucosa sampling

* Able to comprehend the investigational nature of the protocol and provide informed consent (If the healthy volunteer is a minor, the minor s parent or guardian must provide consent and the minor must be able to provide assent)
* Must be willing to allow samples to undergo genetic studies.

EXCLUSION CRITERIA:

* Healthy volunteers and/or pregnant women with diseases with an inflammatory or immune component
* Subjects with active infections requiring systemic antibiotic therapy
* Persons who are alcoholic or abusers of illicit substances

Min Age: 8 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 88 (Actual)
Dates: Start 2009-09-09; Study Completion 2018-09-05

PRIMARY OUTCOMES:
Mechanism for collecting samples | One time point

CONTACTS AND LOCATIONS:
Overall Officials: Angelique Biancotto, Ph.D., Principal Investigator — National Institute of Allergy and Infectious Diseases (NIAID)
Locations (1):
- National Institutes of Health Clinical Center, 9000 Rockville Pike, Bethesda, Maryland, United States